CLINICAL TRIAL: NCT05978830
Title: The Development of Early-stage Alzheimer's Disease Multimodal Fusion Warning System and Non-invasive Neurostimulation Techniques.
Brief Title: Development of Multimodal Fusion Warning System and Non-invasive Techniques for Early Alzheimer's Detection.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diagnosis and prognosis of AD
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer's Disease
Keywords: EEG; MRI; Digital intelligence equipment; Machine learning; microstate
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Cognitive assessment was performed by neuropsychological professionals before and after each treatment, and treatment was performed with real and fake stimuli Multimodal MRI was performed again 2 days later. (1) Subjects in one group received Active Transcranial ultrasound stimulation for 2 weeks ; The other group received Sham Transcranial ultrasound stimulation for 2 weeks.
Who Masked: Participant, Investigator
Masking Description: The study is double-blinded, meaning both participant and Investigator are unaware of the treatment received by the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The group of subjects underwent active Transcranial ultrasound stimulation for 2 weeks
  Interventions: Device: Transcranial ultrasound stimulation
- Group 2 (Sham Comparator): The group of subjects underwent sham Transcranial ultrasound stimulation for 2 weeks
  Interventions: Device: Transcranial ultrasound stimulation

INTERVENTIONS:
Device: Transcranial ultrasound stimulation — In each active/sham-ultrasound stimulation experiment, subjects first underwent two baseline motor evoked potential (MEP) tests, with an interval of 15 minutes between the two baseline tests. After 15 minutes of true/pseudo-transcranial ultrasound stimulation, subjects immediately underwent a MEP test, and then 15 minutes later, subjects underwent another MEP test. The MEP was tested again 15 minutes later.

SUMMARY:
Developing and validating an early digitalized recognition device and multimodal warning model for Alzheimer's disease, and establishing a precision transcranial ultrasound stimulation intervention system.

DETAILED DESCRIPTION:
1. Establishment of early digitalized recognition devices and multimodal warning models for AD: Participants undergo clinical assessments, and if they meet the inclusion criteria, their gender, age, MMSE, MoCA, CDR, GDS scores, as well as EEG ERP and MR data are collected. Eye-tracking analysis based on human-computer interaction perception technology, limb movement detection, and laser radar depth sensor fusion cognitive assessment are also performed simultaneously. After enrollment, follow-up assessments using scales (MMSE, MoCA, CDR, GDS, ADAS-cog, etc.) are conducted every six months, and EEG ERP and MR data are collected annually.
2. Construction of a precision transcranial ultrasound stimulation intervention system: Participants were randomly divided into true stimulation group and false stimulation group: true/false stimulation for 2 weeks, washout for 2 weeks, false/true stimulation for 2 weeks. After treatment, behavioral scale assessment, EEG ERP and multimodal MRI were performed to evaluate the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MCI / AD
2. Between the ages of 55 and 80
3. No history of mental illness such as schizophrenia, severe anxiety and depression

Exclusion Criteria:

1. Consistent with Parkinson's disease, frontotemporal dementia, dementia with lewy bodies Or Huntington's disease diagnostic criteria
2. Dementia due to other causes (e.g. cerebrovascular disease, central nervous system trauma, tumors, infections, Metabolic diseases, normal stress hydrocephalus, folic acid or vitamin B12 deficiency, hypothyroidism, etc.)
3. Have aphasia,Disorders that affect cognitive assessment, such as disorders of consciousness
4. Have a history of epilepsy or take antiepileptic drugs

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Power spectrum | 6 months
  The investigators collected EEG data of participants in resting state and listening to music and the absolute power spectral density values (alpha,beta,theta,delta bands dB/Hz) will be calculated using spectral analysis.
Duration of microstate | 6 months
  The investigators refined the microstate method to accurately estimate topographical differences. The calculations were performed for measures of duration (ms). The duration of each microstate were utilized to predict disease classification and prognosis evaluation for patients with Alzheimer's disease.
Occurrence of microstate | 6 months
  The investigators refined the microstate analysis. The calculations were performed for measures of occurrence (times per minute). The occurrence of microstates were utilized to predict disease classification and prognosis evaluation for patients with disturbance of consciousness.
Mini-Mental State Examination (MMSE) | 6 months
  MMSE includes a series of questions and tasks to assess the individual's memory, attention, calculation, language, spatial, and executive functions. The test items include recalling instructions, reproducing patterns, performing mathematical calculations, naming objects, writing sentences, etc. Each item has different scoring criteria, and scores are assigned based on the participant's responses and performance. The total score is 30, with higher scores indicating better cognitive functioning.
Montreal Cognitive Assessment (MoCA) | 6 months
  MoCA is a standardized assessment tool used to evaluate cognitive function, particularly for early cognitive impairment and mild cognitive impairment. It consists of a series of questions and tasks that cover areas such as memory, attention, executive functions, language, and spatial abilities. Test items include naming animals, drawing a clock, recalling a sequence, task guidance, etc., and each item is assigned a different score. The score range is from 0 to 30, with higher scores indicating better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: benyan luo, Pro, Study Chair — Department of Neurology, First Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Yi Ling, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No